CLINICAL TRIAL: NCT02576522
Title: Tumor Bed Hypofractionated IMRT (VMAT-RA) After Surgical Resection for Patients With Single, Large (≥2.1 cm) Brain Metastases From Solid Tumor
Brief Title: Tumor Bed Hypofractionated IMRT After Surgery for Patients With Single,Large Brain Metastases From Solid Tumor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Principal Investigator, Michele Tedeschi, MD, Istituto Clinico Humanitas
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1408
Record Dates: First submitted 2015-10-07; First posted 2015-10-15 (Estimated); Last update posted 2019-05-28 (Actual); Status verified 2019-05

CONDITIONS: Brain Metastases
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- brain metastatic patients (Experimental): Patients with single, large brain metastases from solid tumors
  Interventions: Radiation: brain metastatic patients

INTERVENTIONS:
Radiation: brain metastatic patients — Surgery followed by hypofractionated intensity modulated radiation therapy (IMRT) using VMAT approach

SUMMARY:
Investigators designed a study of a multimodality approach: surgery followed by hypofractionated intensity modulated radiation therapy (IMRT) using VMAT approach for patients with single, large brain metastases from solid primary tumor

DETAILED DESCRIPTION:
Investigators designed a study to recruit patients with single, large brain metastases from solid primary tumor for a multimodality approach: surgery followed by hypofractionated intensity modulated radiation therapy (IMRT) using VMAT approach. The potential advantage of this treatment is to improve local control and to reduce toxicity compared with WBRT or SRS after surgical resection.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Karnosky performance status (KPS) ≥70
* All Solid tumor (esclusion SCLC and Germinal tumors)
* Controlled primary tumor
* Controlled other metastatic site
* Single metastatic lesion at diagnosis
* Lesions ≥ 2.1 cm in maximum diameter (4 cm3), < 3 cm conditioning mass effect or neurological deficits or massive aedema, unknown primary tumor
* Estimated survival ≥ 3 months.
* Written informed consent

Exclusion Criteria:

* Prior WBRT
* KPS ≤ 70
* Other primary cancer
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2015-06-29 (Actual); Primary Completion 2019-01-22 (Actual); Study Completion 2019-01-22 (Actual)

PRIMARY OUTCOMES:
Local control rate | 6 months

SECONDARY OUTCOMES:
Distant brain failure | 6 months
Overall survival, statistical | 6 months
Morbidity/mortality after surgery | 1 month
Radionecrosis after treatments | 6 months
Neuropsycological alterations after treatments, questionnaire | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Pierina Navarria, MD, Principal Investigator — Istituto Clinico Humanitas
Locations (1):
- Istituto Clinico Humanitas, Rozzano, Milano, Italy